CLINICAL TRIAL: NCT05282836
Title: Early Hydrogen-Oxygen Gas Mixture Inhalation Therapy for Patients With Aneurysmal Subarachnoid Hemorrhage: A Randomized, Controlled Clinical Trial
Brief Title: Early Hydrogen-Oxygen Gas Mixture Inhalation in Patients With Aneurysmal Subarachnoid Hemorrhage (HOMA)
Acronym: HOMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HX-A-2021016
Record Dates: First submitted 2022-03-08; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Nebulizers and Vaporizers

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): H2-O2 (66% hydrogen; 33% oxygen) inhalation. Patients in the treatment group inhaled H2-O2 (66% hydrogen; 33% oxygen) at 3 L/min via nasal cannula by using the Hydrogen/Oxygen Generator (model AMS-H-03, Shanghai Asclepius Meditech Co., Ltd., China) during a 7-day stay in the intensive care unit.
  Interventions: Device: Hydrogen Oxygen Generator with Nebulizer
- No intervention (No Intervention): Usual care refers to the standard-of-care (including oxygen therapy) recommended by guidelines.

INTERVENTIONS:
Device: Hydrogen Oxygen Generator with Nebulizer — Patients in treatment group inhaled H2-O2 (66% hydrogen; 33% oxygen) at 3 L/min via nasal cannula by using the Hydrogen/Oxygen Generator (model AMS-H-03, Shanghai Asclepius Meditech Co., Ltd., China) during a 7-day stay in the intensive care unit.
  Arms: Intervention

SUMMARY:
This was a randomized, single-center trial. On the basis of standard-of-care, patients in the treatment group inhaled H2-O2 (66% hydrogen; 33% oxygen) at 3 L/min via nasal cannula by using the Hydrogen/Oxygen Generator (model AMS-H-03, Shanghai Asclepius Meditech Co., Ltd., China) during a 7-day stay in the intensive care unit. Patients in the control group received standard-of-care (consisting of oxygen therapy) alone. This study intends to apply Hydrogen/Oxygen Generator in clinical patients with aneurysmal subarachnoid hemorrhage (aSAH), exploring the role of hydrogen-oxygen mixed gas inhalation therapy in early brain injury, and the prevention of cerebral vasospasm and delayed cerebral ischemia, finally providing a scientific basis for hydrogen treatment of aSAH.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Signed informed consent
3. Must be admitted within 72 hours after aneurysm rupture

Exclusion Criteria:

1. physical disability caused by any reason before the onset of the disease
2. dementia or mental illness before the onset of the disease
3. more than 72 hours after aneurysm rupture admitted to hospital for treatment
4. do not cooperate with the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2023-03-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
In- hospital Cerebral Vasospasm | From baseline to 14 days
  The proportion of patients with cerebral vasospasm at day 14
In- hospital Delayed Cerebral Ischemia | From baseline to 14 days
  The proportion of patients with delayed cerebral ischemia at day 14

SECONDARY OUTCOMES:
modified Rankin Scale score | 90 days after discharge
  modified Rankin Scale score at 90 days after discharge
Montreal Cognitive Assessment score | 90 days after discharge
  Montreal Cognitive Assessment score at 90 days after discharge

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lin F, Li R, Chen Y, Yang J, Wang K, Jia Y, Han H, Hao Q, Shi G, Wang S, Zhao Y, Chen X. Early Hydrogen-Oxygen Gas Mixture Inhalation in Patients with Aneurysmal Subarachnoid Hemorrhage (HOMA): study protocol for a randomized controlled trial. Trials. 2024 Jun 11;25(1):377. doi: 10.1186/s13063-024-08231-5. PMID 38863026